CLINICAL TRIAL: NCT06774404
Title: Flash Glucose Monitoring Targets in Gestational Diabetes
Acronym: FlaG-TaG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-449/2021/15
Record Dates: First submitted 2024-12-04; First posted 2025-01-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-10

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational diabetes mellitus; Flash Glucose Monitoring; Pregnancy; FGM
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pregnant women with GDM using FGM and SMBG (Experimental): Pregnant women with GDM using Flash Glucose Monitoring (FGM) and Self-Monitoring of Blood Glucose (SMBG)
  Interventions: Device: Use of FreeStyle Libre 14 day Flash Glucose Monitoring System
- Pregnant women with GDM using only SMBG (Active Comparator)
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Use of FreeStyle Libre 14 day Flash Glucose Monitoring System — Women with GDM in the intervention arm will use Flash Glucose Monitoring (FGM) from diagnosis until the end of pregnancy
  Arms: Pregnant women with GDM using FGM and SMBG
Other: No intervention — Only using SMBG
  Arms: Pregnant women with GDM using only SMBG

SUMMARY:
The use of glucose monitoring sensors is already well-established in pregnant women with type 1 diabetes (T1D), where it has been proven to improve glycemic control and perinatal outcomes. However, it has not yet been sufficiently researched in the area of gestational diabetes (GDM). Some smaller studies have shown a favorable effect on glycemic control, but no statistically significant differences were observed in reducing perinatal complications. A randomized, prospective study will include 200 pregnant women with GDM, treated at the Diabetes Outpatient Clinic of the Clinical Department of Endocrinology, Diabetes, and Metabolic Diseases at the University Medical Centre Ljubljana. Participants will be divided into two groups. The first group will measure subcutaneous glucose using FSL in addition to self-monitoring of blood glucose (SMBG) while fasting and 60 minutes after main meals at the same time intervals. In both groups, glycemic targets, maternal outcomes, and neonatal outcomes will be monitored. In the FSL + SMBG group, sensor parameters for glycemic control will also be tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women treated at the Diabetes Outpatient Clinic of the Clinical Department of Endocrinology, Diabetes, and Metabolic Diseases for gestational diabetes (GDM),
2. Agreement with the study protocol and ability to follow the study protocol,
3. Diagnosis of GDM established using the standard recommended OGTT method between the 24th and 28th weeks of pregnancy,
4. Age between 18 and 40 years.

Exclusion Criteria:

1. History of bariatric surgery,
2. Treatment with systemic corticosteroids for more than 14 days prior to inclusion in the study,
3. Multiple pregnancy,
4. Hospitalization for psychiatric illness within the last year,
5. First visit to the Diabetes Outpatient Clinic after the 34th week of gestation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 205 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Up to delivery
  Average Fasting Glucose Concentration: Measured in mmol/L, calculated from fasting blood glucose readings and average Postprandial Glucose Concentration: Measured in mmol/L, based on glucose readings taken 60 minutes after main meals.

SECONDARY OUTCOMES:
Mean Glucose (MG) in FSL+ SMBG group | Up to delivery
  Measured in millimoles per liter (mmol/L), reflecting the average glucose level recorded by the sensor.
Mean Amplitude of Glycemic Excursions (MAGE) (FSL+SMBG group) | Up to delivery
  Measured in millimoles per liter (mmol/L), representing glycemic variability.
Time in Range - TIR (SMBG+FSL group) | Up to delivery
  Defined as the percentage (%) of time sensor glucose levels fall between 3,5 and 7,8 mmol/l
Adherence to the Intervention | Up to delivery
  Measured as the percentage (%) of completed prescribed self-monitoring and sensor glucose readings relative to the total number of prescribed measurements.
Gestational Weight Gain (GWG) | Up to delivery
  Measured in kilograms (kg), calculated as the difference between pre-pregnancy weight and the last recorded weight before delivery.
Mode of Delivery | At delivery
  Categorized into vaginal delivery, assisted vaginal delivery, or cesarean section, and reported as percentages (%) for each category.
Occurrence of Hypertensive Disorders | Up to delivery
  Reported as a binary outcome (Yes/No), based on clinical diagnosis during pregnancy.
Birth Weight | At birth of infant
  Measured in grams (g), recorded immediately after delivery
Large-for-Gestational-Age (LGA) Infant | At birth of infant
  Defined as birth weight above the 90th percentile for gestational age, reported as a binary outcome (Yes/No).
Small-for-Gestational-Age (SGA) Infant | At birth of infant
  Defined as birth weight below the 10th percentile for gestational age, reported as a binary outcome (Yes/No).
Gestational Age at Birth | At birth of infant
  Measured in completed weeks, based on the interval from the first day of the last menstrual period or ultrasound-confirmed dating.
Neonatal Hypoglycemia | At birth of infant
  Defined as blood glucose levels below 2.6 mmol/L in the first 48 hours of life, reported as a binary outcome (Yes/No).
Pregnancy loss | <28 days of life
  Miscarriage, stillbirth, neonatal death
Hyperbilirubinemia | Within first 7 days of life
  Treated with phototherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No